CLINICAL TRIAL: NCT00090766
Title: Safety and Pharmacokinetics of Valganciclovir Syrup Formulation in Pediatric Solid Organ Transplant Recipients
Brief Title: A Study of Valcyte (Valganciclovir) Syrup Formulation in Pediatric Solid Organ Transplant Recipients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WV16726
Record Dates: First submitted 2004-09-03; First posted 2004-09-06 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-03

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir

ARMS (3):
- Valganciclovir Age Group <= 2 Years (Experimental): Eligible participants aged <= 2 years received valganciclovir up to maximum of 900 milligrams (mg) once daily oral dose (solution or tablets) from the time of kidney transplantation for up to 100 days post-transplant. Dose = 7 * body surface area (BSA) * creatinine clearance (CrCLS).
  Interventions: Drug: valganciclovir [Valcyte]
- Valganciclovir Age Group >2 to <12 Years (Experimental): Eligible participants aged >2 to <12 years received valganciclovir up to maximum of 900 mg once daily oral dose (solution or tablets) from the time of kidney transplantation for up to 100 days post-transplant. Dose = 7 * BSA * CrCLS.
  Interventions: Drug: valganciclovir [Valcyte]
- Valganciclovir Age Group >= 12 Years (Experimental): Eligible participants aged >= 12 years received valganciclovir up to maximum of 900 mg once daily oral dose (solution or tablets) from the time of kidney transplantation for up to 100 days post-transplant. Dose = 7 * BSA * CrCLS.
  Interventions: Drug: valganciclovir [Valcyte]

INTERVENTIONS:
Drug: valganciclovir [Valcyte] — po daily (dose based on body surface area and CrCL)

SUMMARY:
This study will assess the safety and pharmacokinetics of Valcyte syrup in pediatric solid organ transplant recipients. The anticipated time on study treatment is 3-12 months and the target sample size is less than 100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* patients between 3 months and 16 years of age;
* first solid organ transplant (eg, kidney, liver, heart);
* able to tolerate oral medication;
* females of childbearing potential must agree to utilize an effective method of contraception throughout the study and for 90 days following discontinuation of study drug;
* patients at risk of developing CMV disease (all transplant recipients other than those who are D-R- for CMV).

Exclusion Criteria:

* patients who have previously participated in this study;
* patients who are participating in another clinical trial (except with the approval of the Sponsor);
* severe, uncontrolled diarrhea (more than 5 watery stools per day);
* pregnant or lactating females.

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2004-05; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- United States (6):
  - Los Angeles, California
  - Indianapolis, Indiana
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - New York, New York
  - Salt Lake City, Utah
- Parkville, Australia
- Canada (2):
  - Edmonton, Alberta
  - Winnipeg, Manitoba
- Paris, France
- Berlin, Germany
- Mexico (2):
  - Guadalajara
  - Mexico City
- Spain (2):
  - Madrid
  - Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 63 participants were enrolled in this study conducted from 28 May 2004 to 13 May 2005. The study was conducted at 18 centers in 7 countries.
Pre-assignment Details: Participants were screened within 48 hours prior to transplant surgery (Day 1) and received valganciclovir from Day 1.
Groups:
- Valganciclovir Age Group <= 2 Years: Eligible participants aged <= 2 years received valganciclovir up to maximum of 900 milligrams (mg) once daily oral dose (solution or tablets) from the time of kidney transplantation for up to 100 days post-transplant. Dose was calculated using the algorithm (7 * body surface area [BSA] * creatinine clearance [CrCLS]).
- Valganciclovir Age Group >2 to < 12 Years: Eligible participants aged >2 to < 12 years received valganciclovir up to maximum of 900 mg once daily oral dose (solution or tablets) from the time of kidney transplantation for up to 100 days post-transplant. Dose was calculated using the algorithm (7 * BSA * CrCLS).
- Valganciclovir Age Group >= 12 Years: Eligible participants aged >= 12 years received valganciclovir up to maximum of 900 mg once daily oral dose (solution or tablets) from the time of kidney transplantation for up to 100 days post-transplant. Dose was calculated using the algorithm (7 * BSA * CrCLS).
Period: Overall Study
Arm/Group | Valganciclovir Age Group <= 2 Years | Valganciclovir Age Group >2 to < 12 Years | Valganciclovir Age Group >= 12 Years
Started | 17 | 21 | 25
Completed | 14 | 19 | 22
Not Completed | 3 | 2 | 3
Not completed — Nephrectomy Planned | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Admin | 0 | 2 | 0
Not completed — Lost to Follow-up | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of valganciclovir
Groups:
- Valganciclovir Age Group <= 2 Years: Eligible participants aged <= 2 years received valganciclovir up to maximum of 900 milligrams (mg) once daily oral dose (solution or tablets) from the time of kidney transplantation for up to 100 days post-transplant. Dose was calculated using the algorithm (7 * BSA * CrCLS).
- Total: Total of all reporting groups
Arm/Group | Valganciclovir Age Group <= 2 Years | Valganciclovir Age Group >2 to < 12 Years | Valganciclovir Age Group >= 12 Years | Total
Number analyzed (Participants) | 17 | 21 | 25 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.6 (0.86) | 6.9 (3.15) | 14.2 (1.54) | 8.1 (5.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 13 | 29
  Male | 8 | 14 | 12 | 34

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Concentration-Time Curve From 0 to 24 Hours of Valganciclovir
Description: Area Under the Plasma Concentration-Time Curve (AUC) is a measure of the plasma concentration of the drug over time. The AUC 0-24 hours is area under the plasma concentration-time curve from time zero through 24 hours after dosing. A compartmental model was used to measure the plasma concentrations of valganciclovir. One participant was not analyzed for this outcome measure as the participant underwent both a kidney and liver transplant.
Time Frame: Pre-dose; 1-3, 3-7, 7-12 hours post dose on any day between Day 7 to Day 14; Week 6, Week 10, and Week 14
Population: Pharmacokinetic (PK) population comprised of all participants from studies WP16296, WP16303 and WV16726 who had completed the specified treatment and from whom at least one plasma sample was taken. Here n represents number of participant with specific transplant i.e., kidney, liver, and heart.
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Groups:
- Valganciclovir Age Group <= 2 Years: Eligible participants aged <= 2 years received valganciclovir up to maximum of 900 mg once daily oral dose (solution or tablets) from the time of kidney transplantation for up to 100 days post-transplant. Dose was calculated using the algorithm (7 * BSA * CrCLS).
Arm/Group | Valganciclovir Age Group <= 2 Years | Valganciclovir Age Group >2 to < 12 Years | Valganciclovir Age Group >= 12 Years
Number analyzed (Participants) | 17 | 20 | 25
mcg*hr/mL
  In kidney recipients, n=2, 12, 19 | 65.2 (16.6) | 55 (11.9) | 50 (11.6)
  In liver recipients, n=9, 6, 2 | 69.4 (35.4) | 58.4 (6.18) | 35.6 (2.76)
  In heart recipients, n=6, 2, 4 | 56.3 (23.2) | 60 (19.3) | 61.2 (26)

2. Primary Outcome: Number of Participants With Adverse Events Leading to Dose Interruption or Modification
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation in participant administered a pharmaceutical product, which did not necessarily have to have a causal relationship with this treatment. The number of participants with AEs leading to dose interruptions or modifications are reported.
Time Frame: Up to Week 26
Population: Safety population included all participants who received at least one dose of valganciclovir.
Measure: Number; unit: participants
Groups:
- Valganciclovir Age Group >= 12 Years: Participants aged >= 12 years received a once daily oral dose (solution or tablets) of valganciclovir from the time of kidney transplant for up to 100 days post-transplant. Dose (in mg) was calculated using the algorithm (7 * body surface area * creatinine clearance).
Arm/Group | Valganciclovir Age Group <= 2 Years | Valganciclovir Age Group >2 to < 12 Years | Valganciclovir Age Group >= 12 Years
Number analyzed (Participants) | 17 | 21 | 25
participants | 4 | 2 | 3

3. Primary Outcome: Number of Participants With Opportunistic Infections
Description: Opportunistic infections included oral candidiasis, candidiasis, herpes simplex, cytomegalovirus antigen positive, cytomegalovirus test positive. The number of participants with opportunistic infections are reported.
Time Frame: Up to Week 26
Population: Safety population included all participants who received at least one dose of valganciclovir.
Measure: Number; unit: participants
Arm/Group | Valganciclovir Age Group <= 2 Years | Valganciclovir Age Group >2 to < 12 Years | Valganciclovir Age Group >= 12 Years
Number analyzed (Participants) | 17 | 21 | 25
participants
  Oral Candidiasis | 2 | 0 | 0
  Candidiasis | 1 | 0 | 0
  Herpes Simplex | 0 | 1 | 0
  Cytomegalovirus Antigen Positive | 1 | 0 | 0
  Cytomegalovirus Test Positive | 1 | 0 | 0

4. Primary Outcome: Number of Participants With Any Adverse Events and Any Serious Adverse Events
Description: An AE was defined as any untoward medical occurrence in a clinical investigation in participant administered a pharmaceutical product, which did not necessarily have to have a causal relationship with this treatment. A serious adverse event (SAE) is any experience or a significant hazard, that is fatal, life-threatening, requires in-patient hospitalization or prolongation of existing one, results in persistent or significant disability, is a congenital anomaly, is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: Up to Week 26
Population: Safety population included all participants who received at least one dose of valganciclovir.
Measure: Number; unit: participants
Arm/Group | Valganciclovir Age Group <= 2 Years | Valganciclovir Age Group >2 to < 12 Years | Valganciclovir Age Group >= 12 Years
Number analyzed (Participants) | 17 | 21 | 25
participants
  Any AE | 17 | 18 | 24
  Any SAE | 13 | 11 | 11

5. Primary Outcome: Number of Participants With Adverse Events Leading to Discontinuation of the Study Drug
Description: An AE was defined as any untoward medical occurrence in a clinical investigation in participant administered a pharmaceutical product, which did not necessarily have to have a causal relationship with this treatment. The number of participants with AEs leading to discontinuation of the study drug is reported.
Time Frame: Up to Week 26
Population: Safety population included all participants who received at least one dose of valganciclovir.
Measure: Number; unit: participants
Arm/Group | Valganciclovir Age Group <= 2 Years | Valganciclovir Age Group >2 to < 12 Years | Valganciclovir Age Group >= 12 Years
Number analyzed (Participants) | 17 | 21 | 25
participants | 1 | 2 | 0

6. Primary Outcome: Number of Participants With 3 Grade Shift From Baseline of Adverse Events in Hematology and Serum Chemistry
Description: The number of participants experiencing a 3 grade shift (example from Grade 0 to Grade 3) from baseline (BL) in hematology and serum chemistry laboratory parameters are reported. The data was analyzed for overall study only.
Time Frame: Up to Week 26
Population: Safety population included all participants who received at least one dose of valganciclovir.
Measure: Number; unit: participants
Groups:
- Overall Study: All participants who received at least one dose of valganciclovir up to maximum of 900 mg once daily oral dose (solution or tablets) from the time of kidney transplantation for up to 100 days post-transplant. Dose was calculated using the algorithm (7 * BSA * CrCLS).
Arm/Group | Overall Study
Number analyzed (Participants) | 63
participants
  Hemoglobin low, n= 63 | 6
  White blood cell count low, n= 59 | 3
  Lymphocytes low, n= 54 | 3
  Neutrophils low, n= 54 | 7
  Potassium low, n=56 | 4
  Potassium high, n=57 | 4
  Alkaline Phosphatase high, n=40 | 1
  Alanine transaminase high, n=48 | 1
  Total Bilirubin high, n=38 | 1
  Sodium low, n=58 | 2
  Sodium high, n=57 | 0
  Calcium low, n=46 | 1
  Phosphate low, n=43 | 2
  Fasting Glucose low, n=39 | 1
  Uric Acid high, n=21 | 2

7. Primary Outcome: Number of Participants With 4 Grade Shift From Baseline of Adverse Events in Hematology and Serum Chemistry
Description: The number of participants experiencing a 4 grade shift (example from Grade 0 to Grade 4) from BL in hematology and serum chemistry laboratory parameters are reported. The data was analyzed for overall study only.
Time Frame: Up to Week 26
Population: Safety population included all participants who received at least one dose of valganciclovir.
Measure: Number; unit: participants
Arm/Group | Overall Study
Number analyzed (Participants) | 63
participants
  Hemoglobin low, n= 63 | 0
  White blood cell count low, n= 59 | 1
  Lymphocytes low, n= 54 | 3
  Neutrophils low, n= 54 | 4
  Potassium low, n=56 | 0
  Potassium high, n=57 | 2
  Alkaline Phosphatase high, n=40 | 0
  Alanine transaminase high, n=48 | 0
  Total Bilirubin high, n=38 | 0
  Sodium low, n=58 | 0
  Sodium high, n=57 | 1
  Calcium low, n=46 | 3
  Phosphate low, n=43 | 0
  Fasting Glucose low, n=39 | 0
  Uric Acid high, n=21 | 2

8. Secondary Outcome: Number of Participants With Cytomegalovirus Disease Over Time
Description: Cytomegalovirus (CMV) disease is defined as syndrome or tissue invasive disease in which CMV virus was identified in blood, urine, biopsy or other suitable specimen, which could be in conjunction with one or more of the following events: a) CMV syndrome was defined as virus present in blood or other suitable specimen, plus fever, and any of the following: leukopenia, atypical lymphocytosis, thrombopenia or elevated hepatic transaminases (for non-liver recipients). b) The diagnosis of organ specific tissue invasive CMV disease was evidence of CMV in the tissue (CMV inclusion bodies or in situ detection of CMV antigen or DNA), plus signs/symptoms of organ dysfunction.
Time Frame: Up to Week 26
Population: Safety population included all participants who received at least one dose of valganciclovir.
Measure: Number; unit: participants
Arm/Group | Valganciclovir Age Group <= 2 Years | Valganciclovir Age Group >2 to < 12 Years | Valganciclovir Age Group >= 12 Years
Number analyzed (Participants) | 17 | 21 | 25
participants | 0 | 2 | 2

9. Secondary Outcome: Number of Participants With Treatment Failures
Description: Treatment failure was defined as either the development of CMV (viremia, antigenemia or test positive) requiring treatment up to day 100 post-transplant (i.e, while undergoing prophylaxis with valganciclovir up to day 100) or discontinuation of study medication due to lack of efficacy or to toxicity.
Time Frame: Up to Week 26
Population: The Intent to Treat (ITT) population comprised all participants who received at least one dose of the study drug, whether on-study or prematurely withdrawn.
Measure: Number; unit: participants
Arm/Group | Valganciclovir Age Group <= 2 Years | Valganciclovir Age Group >2 to < 12 Years | Valganciclovir Age Group >= 12 Years
Number analyzed (Participants) | 17 | 21 | 25
participants | 2 | 2 | 0

10. Secondary Outcome: Number of Participants Who Experienced Graft Loss
Description: Graft loss was defined as impairment of organ function to such a degree that the participant died or underwent re-transplantation.
Time Frame: Up to Week 26
Population: ITT population: The ITT population comprised all participants who received at least one dose of the study drug, whether on-study or prematurely withdrawn.
Measure: Number; unit: participants
Arm/Group | Valganciclovir Age Group <= 2 Years | Valganciclovir Age Group >2 to < 12 Years | Valganciclovir Age Group >= 12 Years
Number analyzed (Participants) | 17 | 21 | 25
participants
  Acute Graft Rejection | 1 | 0 | 0
  Chronic Graft Rejection | 0 | 0 | 0
  Recurrence of Underlying Disease | 0 | 0 | 0
  Technical Complications | 0 | 0 | 1
  Primary Graft Non-Function | 0 | 0 | 0
  Other | 0 | 1 | 0

11. Secondary Outcome: Mean Maximum Plasma Concentration of Valganciclovir Over Time
Description: Maximum Plasma Concentration (Cmax) is defined as the maximum observed plasma concentration of Valganciclovir. Participants with kidney, liver and heart transplant were analyzed. One participant was not analyzed for this outcome measure as the participant underwent both a kidney and liver transplant.
Time Frame: Pre-dose; 1-3, 3-7, 7-12 hours post dose on any day between Day (D) 7 to D 14; and at Week (W) 6, W 10, and W 14
Population: The PK analysis population comprised all participants from studies WP16296, WP16303 and WV16726 who completed the specified treatment and from whom at least one plasma sample was taken. Here n represents number of participant with specific transplant i.e., kidney, liver, and heart.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Valganciclovir Age Group <= 2 Years | Valganciclovir Age Group >2 to < 12 Years | Valganciclovir Age Group >= 12 Years
Number analyzed (Participants) | 17 | 20 | 25
mcg/mL
  In kidney recipients, n=2, 12, 19 | 10 (0.04) | 8.74 (2.49) | 7.85 (2.1)
  In liver recipients, n=9, 6, 2 | 11.7 (3.59) | 9.35 (2.33) | 5.55 (1.34)
  In heart recipients, n=6, 2, 4 | 8.22 (2.44) | 12.5 (1.02) | 9.5 (3.34)

12. Secondary Outcome: Mean Elimination Half-Life of Valganciclovir Over Time
Description: The Elimination Half-Life Period is defined as the time measured for the plasma concentration to decrease by half to its original concentration. One participant was not analyzed for this outcome measure as the participant underwent both a kidney and liver transplant. Here n represents number of participant with specific transplant i.e., kidney, liver, and heart.
Time Frame: Pre-dose; 1-3, 3-7, 7-12 hours post dose on any day between Day 7 to Day 14; Week 6, Week 10, and Week 14
Population: The PK analysis population comprised all participants from studies WP16296, WP16303 and WV16726 who completed the specified treatment and from whom at least one plasma sample was taken.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Valganciclovir Age Group <= 2 Years | Valganciclovir Age Group >2 to < 12 Years | Valganciclovir Age Group >= 12 Years
Number analyzed (Participants) | 17 | 20 | 25
hours
  In kidney recipients, n=2, 12, 19 | 3.1 (0.59) | 4.47 (1.37) | 5.69 (1.06)
  In liver recipients, n=9, 6, 2 | 2.72 (1.32) | 3.61 (0.8) | 4.5 (0.25)
  In heart recipients, n=6, 2, 4 | 3.6 (1.73) | 2.62 (0.65) | 5.05 (0.7)

13. Secondary Outcome: Number of Participants Who Experienced Episodes of Rejection Over Time
Description: Participants with biopsy proven active rejection are reported.
Time Frame: Up to Week 26
Population: The ITT population comprised all participants who received at least one dose of the study drug, whether on-study or prematurely withdrawn.
Measure: Number; unit: participants
Arm/Group | Valganciclovir Age Group <= 2 Years | Valganciclovir Age Group >2 to < 12 Years | Valganciclovir Age Group >= 12 Years
Number analyzed (Participants) | 17 | 21 | 25
participants | 5 | 2 | 2

ADVERSE EVENTS:
Time Frame: Up to Week 26
Description: Serious adverse events and non-serious adverse events are reported in safety analysis set, which consists of all participants who received at least one dose of study drug and had a safety assessment performed post baseline.
Arm/Group | Valganciclovir Age Group <= 2 Years | Valganciclovir Age Group >2 to < 12 Years | Valganciclovir Age Group >= 12 Years
Serious Adverse Events (participants affected / at risk) | 13/17 | 11/21 | 11/25
Other Adverse Events (participants affected / at risk) | 17/17 | 17/21 | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valganciclovir Age Group <= 2 Years (N=17) | Valganciclovir Age Group >2 to < 12 Years (N=21) | Valganciclovir Age Group >= 12 Years (N=25)
Haematoma (Vascular disorders) | 0 | 1 | 0
Lymphocele (Vascular disorders) | 0 | 0 | 1
Gastrostomy tube insertion (Surgical and medical procedures) | 0 | 1 | 0
Plasmablastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Transplant rejection (Immune system disorders) | 1 | 0 | 3
Pyrexia (General disorders) | 1 | 2 | 1
Chest pain (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cytomegalovirus test positive (Investigations) | 1 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0
Cytomegalovirus antigen positive (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Leukoencephalopathy (Nervous system disorders) | 1 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Hepatic artery thrombosis (Hepatobiliary disorders) | 1 | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic artery stenosis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1 | 0
Cytomegalovirus Viraemia (Infections and infestations) | 0 | 2 | 1
Epstein-barr virus infectionn (Infections and infestations) | 1 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0
Biliary tract infection (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valganciclovir Age Group <= 2 Years (N=17) | Valganciclovir Age Group >2 to < 12 Years (N=21) | Valganciclovir Age Group >= 12 Years (N=25)
Hypertension (Vascular disorders) | 4 | 6 | 8
Haematoma (Vascular disorders) | 1 | 0 | 0
Liver Transplant Rejection (Immune system disorders) | 2 | 0 | 0
Transplant Rejection (Immune system disorders) | 2 | 0 | 0
Milk Allergy (Immune system disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 5 | 8 | 4
Oedema Peripheral (General disorders) | 0 | 0 | 5
Irritability (General disorders) | 2 | 0 | 0
Catheter Site Discharge (General disorders) | 1 | 0 | 0
Catheter Site Inflammation (General disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Incision site infection (Injury, poisoning and procedural complications) | 0 | 2 | 4
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 1
Device Failure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Graft Ischaemia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative Thoracic procedure complications (Injury, poisoning and procedural complications) | 1 | 0 | 0
Epstein-Barr Virus Test positive (Investigations) | 0 | 2 | 0
Blood Albumin Decreased (Investigations) | 1 | 0 | 0
White Blood Cell Count Increased (Investigations) | 1 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1 | 2
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac Disorder (Cardiac disorders) | 1 | 0 | 0
Left Ventricular Failure (Cardiac disorders) | 1 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 9 | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 3 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Thrombocythaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 4
Convulsion (Nervous system disorders) | 2 | 1 | 0
Dystonia (Nervous system disorders) | 1 | 0 | 0
Encephalomalacia (Nervous system disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 8 | 6
Vomiting (Gastrointestinal disorders) | 2 | 7 | 7
Nausea (Gastrointestinal disorders) | 0 | 2 | 6
Constipation (Gastrointestinal disorders) | 0 | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 1
Abdominal Distention (Gastrointestinal disorders) | 0 | 2 | 1
Ascites (Gastrointestinal disorders) | 3 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Teething (Gastrointestinal disorders) | 1 | 0 | 0
Biliary Tract Disorder (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 4 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 2
Acute Prerenal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 4 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 4 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Feeding disorder (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Upper Respiratory Tract (Infections and infestations) | 4 | 5 | 7
Nasopharyngitis (Infections and infestations) | 1 | 1 | 3
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 4
Otitis Media (Infections and infestations) | 1 | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 1
Clostridium Colitis (Infections and infestations) | 1 | 0 | 1
Epstein-Barr Virus Infection (Infections and infestations) | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0
Oral Candidiasis (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 2 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0
Abdominal Infection (Infections and infestations) | 1 | 0 | 0
Candidiasis (Infections and infestations) | 1 | 0 | 0
Central Line Infection (Infections and infestations) | 1 | 0 | 0
Para Influenzae Virus Infection (Infections and infestations) | 1 | 0 | 0
Pneumonia Bacterial (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Stenotrophomonas infection (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.